| Official | Title: Exploring the impact of scaling up mass testing, treatment and tracking on malaria |
|---|---|
| prevalence among children in the Pakro sub district of Ghana | |

NCT:

**Date:** 30/03/2019

**Document:** Study Results

## Coverage

Four MTTT interventions were conducted in July 2017, November 2017, March 2018 and July 2018. Of the 5,000 participants initially targeted across communities for each intervention, coverage ranged from 77.8% (3891/5000) to 98.8% (4,941/5,000) (Table 1). A total of 2,669 participants received all four MTTTs (53%) and the median number of MTTTs participants received was 3. The proportions represent those who were effectively reached and tested. Females made up 50.4% and 52.4% of participants in July 2017 and July 2018, respectively (Table 1).

## Asymptomatic parasitaemia prevalence

Table 1: Parasite carriage across different communities at different time points in the Pakro sub-district

## Prevalence of asymptomatic parasitaemia among community members N (%)

| Characteristics | July 2017 Survey<br>n/N (%) | November 2017<br>Survey n/N (%) | March 2018<br>Survey n/N (%) | July 2018 Survey<br>n/N (%) |
|---|---|---|---|---|
| Community | | | | |
| Abease | 282/888 (31.8) | 124/712 (17.4) | 77/709 (10.9) | 161/721 (22.3) |
| Adesa | 158/406 (38.9) | 85/323 (26.3) | 62/351 (17.7) | 121/342 (35.4) |
| Adjanase | 514/1342 (38.3) | 191/957 (20.0) | 283/1070 (26.5) | 387/1037 (37.3) |
| Fante Town | 543/1530 (35.5) | 306/1238 (24.7) | 347/1284 (27.0) | 392/1236 (31.7) |
| Odumtokro | 101/245 (41.2) | 42/213 (19.7) | 43/190 (22.6) | 63/180 (35.0) |
| Piem | 80/220 (36.4) | 35/183 (19.3) | 50/157 (31.9) | 57/160 (35.6) |
| Sachi/Tabankro | 117/310 (37.7) | 75/265 (28.3) | 75/277 (27.1) | 122/290 (42.1) |
| Total | 1795/4941 (36.3) | 858/3891 (22.1) | 937/4038 (23.2) | 1303/3966 (32.9) |
| Coverage | 4941/5000(98.8) | 3891/5000(77.8) | 4038/5000(80.8) | 3966/5000 (79.3) |

An increase in parasite carriage was observed for Sachi/Tabankro from July 2017 to July 2018. However, this was not significant, (Table 2).

The highest decline in parasitaemia carriage, was observed in Abease while the lowest decline was observed in Adesa. It is not clear what accounted for the heterogeneity as there were no other interventions in the area at the time of this study. Asymptomatic parasitaemia prevalence from July 2017 and July 2018

significantly decreased in both children and adults (p=0.002 for <15 children and p=0.001 for ≥15 years) (Table 2).

As per age group, asymptomatic parasitaemia prevalence significantly declined in the age groups 5-14 and 15-45 years, but the decline was marginally significant in the age group 1-4. This decline in parasitaemia was not significant in the age groups 46-65 and >65 years. An increase in parasitaemia prevalence was observed among the <1 year old age group between July 2017 and 2018. But this was not significant.

Table 2: Univariate analysis of effect of MTTT interventions on prevalence of asymptomatic malaria parasitaemia over the time points July 2017 and 2018.

| Characteristics | July 2017 Survey | July 2018 Survey | $\chi^2$ value | P value |
|---|---|---|---|---|
| Community | n/N (%) | n/N (%) | | |
| Abease | 282/888 (31.8) | 161/721 (22.3) | 17.1 | <0.001** |
| Adesa | 158/406 (38.9) | 121/342 (35.4) | 1 | 0.319 |
| Adjanase | 514/1342 (38.3) | 387/1037 (37.3) | 0.2 | 0.624 |
| Fante Town | 543/1530 (35.5) | 392/1236 (31.7) | 4.4 | 0.037** |
| Odomtokro | 101/245 (41.2) | 63/180 (35.0) | 1.7 | 0.193 |
| Piem | 80/220 (36.4) | 57/160 (35.6) | 0 | 0.882 |
| Sachi/Tabankro | 117/310 (37.7) | 122/290 (42.1) | 1.17 | 0.279 |
| All Communities | 1795 (36.3) | 1303 (32.9) | 11.71 | 0.001** |
| Age_group (years) | n/N (%) | n/N (%) | | _ |
| 0 - 11 months | 14/56 (25.0) | 22/57 (38.6) | 2.4 | 0.121 |
| 1 - 4 years | 270/541 (49.9) | 216/491 (44.0) | 3.6 | 0.057 |
| 5 - 14 years | 759/1387 (54.7) | 582/1180 (49.3) | 7.5 | 0.006** |
| 15 - 45 years | 5852092 (28.0) | 360/1523 (23.6) | 8.5 | 0.003** |
| 46 - 65 years | 129/640 (20.2) | 97/544 (17.8) | 1 | 0.310 |
| > 65 years | 38/225 (16.9) | 26/171 (15.2) | 0.2 | 0.352 |
| Total # of <15 | 1043/1984 (52.6) | 820/1728 (47.5) | 9.7 | 0.002** |
| Total # of ≥15 | 752/2957 (25.4) | 483/2238 (21.6) | 10.4 | 0.001** |
| Mean axillary | | | | |
| Temperature | 36.0 | 36.2 | | <0.001** |
| Use ITN | | | | |
| No | 1595/4574 (34.9) | 380/1166 (32.5) | 0.0012 | <0.001 |
| Yes | 200/367 (54.5) | 923/2800 (33.0) | | |

<sup>\*\*</sup> Significance level at  $\alpha$  =0.05